CLINICAL TRIAL: NCT00876070
Title: Community Oncology Setting Cost Analysis and Disease Outcomes of Taxane Use in Metastatic Breast Cancer
Status: Completed | Type: Observational
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: SCRI OUTCOMES 02
Record Dates: First submitted 2009-04-02; First posted 2009-04-06 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-11

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer; Breast Cancer; MBC; Abraxane; Paclitaxel; Taxol; Docetaxel; Taxotere
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective medical record abstraction study. It is a review and evaluation of up to 300 metastatic breast cancer patients treated with Abraxane or other taxanes such as paclitaxel and docetaxel to determine the overall cost of care for Abraxane compared to other taxanes in the first-line metastatic cancer setting and the cost of care for Abraxane compared to other taxanes when broken down by individual components of cost. In addition, the investigators will review the following patient outcomes: response rate, duration of therapy, toxicity, and survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have received Abraxane chemotherapy greater than three months from the time of chart review.
* Patients that have received taxane chemotherapy greater than three months from the time of chart review.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Metastatic Breast Cancer from January 2005 to three months prior to site-specific protocol initiation will be eligible. This will include current/actively being treated patients as well as patients who have previously completed therapy.
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2008-11; Primary Completion 2009-11 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Describe patient demographics, disease and treatment characteristics. | 6 months

SECONDARY OUTCOMES:
Describe detailed treatment and response characteristics. | 6 months
Describe resource utilization and cost variables. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey F Patton, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (2):
- United States (2):
  - Georgia Cancer Specialists, Atlanta, Georgia
  - Tennessee Oncology, PLLC, Nashville, Tennessee